CLINICAL TRIAL: NCT05509504
Title: A Feasibility Study of Low-Intensity Online Intervention (LiON) for Distressed Youths in Hong Kong
Brief Title: Low-intensity Online Intervention for Young People (Service)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Yi-Nam Suen, Research Assistant Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LiON
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Distress, Emotional

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Low-intensity online intervention
- Control (No Intervention)

INTERVENTIONS:
Other: Low-intensity online intervention — The LiON in the current study is comprised of three core modules identified to be core areas of stress and needs of participants based on clinical experiences of the research team. The three modules include (1) stress management, (2) sleep and relaxation, and (3) problem-solving skills. Each module consists of four 1-on-1 sessions which will be conducted through online platforms (such as Zoom) that lasts for ~45 minutes. Participants will attend these sessions once a week.
  Arms: Intervention

SUMMARY:
Studies have found up to 75% of mental disorders in adulthood have their onset before the age of 25 (Lin et al., 2008; Kessler et al., 2005), suggesting youth marks a critical period of intervention. Across the various psychiatric conditions, depressive and anxiety disorders have consistently been reported to be two of the most common conditions in young people globally (Merikangas et al., 2010; Racine et al., 2021).

Both depressive and anxiety disorders are related to various negative impacts on youths' lives, such as undermining academic achievements, with other negative influences found in past studies (Birmaher et al., 1996; Fletcher, 2008, Woodward and Fergusson, 2001; Swan and Kendall, 2016). Notably, an increasing number of studies have found not only can clinical disorders, but also early symptoms of such conditions, can cause significant burden on the individual, their family and peers, as well as the larger society (Spencer et al., 2018; Lynch and Clarke, 2006; Wingrove and Rickwood, 2020).

Existing healthcare services, however, tend to prioritise service targeting those with severe mental health needs. Knowledge about subtle mental health symptoms is lacking among the general public, which can contribute to delayed care and treatment (Fung et al., 2021). In addition, mental health services in Hong Kong are not only characterised by long waiting times but are also coupled with significant stigma, which can in turn prevent help-seeking, especially among young people (Sun et al., 2017; Yap, Wright, and Jorm, 2011). In view of the significance of early engagement and intervention for those with mental health needs and the current situation in Hong Kong, the implementation of low-intensity online-based interventions (LiON) for mental health appears to be a largely promising approach.

Low-intensity refers to low usage of "specialist therapist time" (Bower and Gilbody, 2005), or usage in a cost-effective way, such as in a group-based Cognitive Behavioural Therapy context. Low-intensity interventions focus on delivering self-help and self-management skills which can be led by non-specialists, which in turn help to reduce the cost required in both training and the delivering of intervention. Recent studies have also increasingly highlighted young people's preference to access mental health services through online platforms (Becker et al., 2016). Due to limited mental health resources and the high demand for mental health services in Hong Kong, such online-based low-intensity interventions - when shown to be effective - can be largely helpful in reducing societal costs, reduce the barriers to help-seeking, and facilitate large-scale implementation of mental health services on a population level.

This study will adopt an open labelled non-randomised controlled design. Participants will be youths receiving low-intensity online intervention (LiON) group or community youths who had no intervention.

The LiON intervention group will first receive the 4-week LiON, with generic self-help tips provided to each participant before completing the T2 assessment.

Prior to the commencement of the LiON, all participants will first be screened for eligibility for participation by a professional clinician of the research team (i.e., psychiatrists or psychologist, senior social worker). A review session via Zoom will also be first provided by the trained interventionist (who will be a graduate with background in psychology, social work, or other related mental health disciplines with prior and ongoing training from senior clinicians of the research team) to each participant to determine his or her needs and ensure all inclusion and exclusion criteria are met. Briefing about the LiON, such as module structure and components of focus will also be provided during this session.

ELIGIBILITY:
Inclusion Criteria:

* young people aged between 12-30
* who have sufficient proficiency in Chinese to understand verbal and written instructions and give informed consent

Exclusion Criteria:

* receiving any form of cognitive behavioural therapy (CBT)
* active suicidal ideation/attempts, serious suicidal ideation or self harm risks within the past one month
* inability to turn on camera for the course of the LiON intervention
* inability to provide emergency contact
* located outside of Hong Kong

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Symptoms of distress | Immediate post-intervention
  6 items from the Kessler Kessler Psychological Distress Scale (K6). The scores range from 0 - 24. Higher scores indicate greater distress level.

SECONDARY OUTCOMES:
Perceived sleep quality | Immediate post-intervention
  1 item from the Pittsburgh Sleep Quality Index (PSQI). The scores range from 1 - 4. Higher scores indicate poorer sleep quality.
Stress coping abilities | Immediate post-intervention
  Brief Resilience Scale (BRS). The scores range from 6-30. Higher scores indicate lower level of resilience.
General self-efficacy | Immediate post-intervention
  General Self-Efficacy Scale (GSE). The scores range from 2-8. Higher scores indicate lower level of self-efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong